CLINICAL TRIAL: NCT03599843
Title: Activating Cancer Communities Through an Exercise Strategy for Survivors (ACCESS)
Brief Title: Activating Cancer Communities Through an Exercise Strategy for Survivors
Acronym: ACCESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1023682
Record Dates: First submitted 2018-07-03; First posted 2018-07-26 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Type 2, hybrid implementation-effectiveness study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ACCESS (Experimental): Individuals that consent to the study will be assigned to a 12-week exercise program (ACCESS)
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Participants will complete a 12 week exercise session that will be comprised of aerobic and/or resistance and/or flexibility training.

SUMMARY:
Cancer continues to have the dubious honor of being the leading cause of premature mortality in Canada. The good news is, advances in early detection and cancer treatments are extending the lives of those diagnosed with the disease. However, as more people are living longer, the impact of the therapies used to treat the disease are becoming increasingly apparent. Ranging from the physiological to psychological, cancer survivors are often confronted with substantial, disabling, and life-threatening consequences. The benefits of physical activity (all movement) and exercise more specifically have long been established as a means of prevention and treatment of chronic disease. Several recent reviews and meta-analyses have demonstrated that exercise is a safe and effective means of preventing and improving a multitude of physical and psychological treatment and disease-related sequelae across the cancer trajectory. For example, we know that cancer survivors who exercise not only have a reduced risk of disease recurrence and cancer mortality, but also have reduced acute/late effects of their cancer and/or its treatment such as anxiety, depression, and cancer-related pain. Regrettably, despite our substantial knowledge base, the majority of cancer survivors are not sufficiently active to realize these benefits over the long-term. Moreover, even with the development of evidence-based guidelines, exercise has not yet been widely implemented as a standard of care in the oncology setting largely due to a lack of resources, exercise expertise, and awareness of benefits. Continuing to provide cancer care with little guidance and understanding of the benefits of exercise places cancer survivors at an increased risk for recurrence, late effects, and/or onset of additional co-morbidities, and premature mortality. Therefore, it is important to consider best practices that will optimize and improve quality of survival. Building on the ongoing work of our Alberta-based colleagues and the Alberta Cancer Exercise (ACE) Program (an evidence-based clinic-to-community cancer exercise model), Activating Cancer Communities through an Exercise Strategy for Survivors (ACCESS) is designed to bridge the gap between research and practice and in doing so, lessen the impact of a cancer diagnosis and its treatment(s) on the physical and psychological well-being of cancer survivors.

DETAILED DESCRIPTION:
Study Design: Type 2, hybrid implementation-effectiveness study The proposed project is strongly aligned with the multidisciplinary Alberta Cancer Exercise (ACE; Culos-Reed and McNeely, Co-PIs) lifestyle initiative - a result of the accumulation of over 15 years of research in the design, implementation and evaluation of cancer exercise programs. While the Alberta model has and will continue to be adapted to the Nova Scotia context, the utilization of a Canadian-based, integrated cancer exercise model, with demonstrated success and existing training resources will provide the much-needed framework to improve health outcomes in cancer patients/survivors. In brief, ACCESS will facilitate oncologist referral of survivors to a hospital-based, Certified Exercise Physiologist (CEP) as well as "Cancer Exercise Wise" certified community-based fitness professionals. The CEP will be responsible for screening and triaging survivors to assess participant interests and needs and to determine the appropriate level of activity and any supervision required to maximize benefits and ensure participant safety. Following screening the CEP will link the survivor with the appropriate hospital or community-based physical activity supports (see "TRIAGE PATHWAY"). Exercise programming will include aerobic, resistance, balance, and flexibility training and will be consistent with the exercise delivery model developed for ACE (www.albertacancerexercise.com). Participants will include adult cancer survivors of all cancers and stages at any point along the cancer care trajectory. Eligibility: Participants will be screened for eligibility and must: 1) Have a diagnosis of cancer; 2) Be 18+ years; 3) Be able to participate in mild levels of physical activity (at a minimum); 4) Be pre-treatment, receiving active treatment, or have received cancer treatment within the past 5 years or have a late presenting/ongoing side-effects related to the cancer diagnosis; 5) be willing to attend a 12-week exercise program in Halifax; and 5) Be able to provide informed written consent in English. A Certified Exercise Physiologist (CEP), housed within the QEII cancer care center (Halifax, NS), will have (medically approved) consenting participants complete a baseline PA and cancer specific screening measure to determine appropriateness/preferences for hospital and/or community-based PA participation. The CEP will oversee baseline physical fitness testing and will evaluate screening and testing results. The CEP will then triage the participant to a hospital or a local community-based fitness center depending on their cancer-related needs and programming preferences. The hospital site, under direct supervision of the CEP, will be used for those with identified cancer or other health-related needs that preclude exercising in a community-based setting. The community-based site will be supported by the CEP and will serve those participants cleared to exercise under a "Cancer and Exercise" trained fitness professional, but without high medical needs that would require direct CEP supervision. INTERVENTION: PA programming will be consistent with the exercise delivery models used in pilot programming both in Alberta and here in Halifax (EXACT) and will include a combination of aerobic, resistance, balance, and flexibility exercises delivered in a circuit-type class setting or group/individual personal training format, twice weekly, for 12-weeks. OUTCOME MEASURES: A mixed-methods approach will be used to assess study outcomes. Patient reported outcomes (effectiveness measures) will be assessed at baseline, post-intervention, 6 and 12 month follow-up. Implementation outcomes will be assessed throughout the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of cancer;
* Be 18+ years;
* Be pre-treatment, receiving active treatment, or have received cancer treatment within the past 5 years or have a late presenting/ongoing side-effects related to the cancer diagnosis;
* Be able to participate in mild levels of physical activity (at a minimum);
* Be willing to attend a 12-week exercise program in Halifax;
* Be able to provide informed written consent in English.

Exclusion Criteria:

- Less than 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Physiological Outcome - resting heart rate | 12 weeks
  Seated resting heart rate will be measured in beats per minute.
Physiological outcome - blood pressure | 12 weeks
  Seated systolic and diastolic blood pressure will be measured in mm of Hg
Physiological outcome - 6 minute walk test (6MWT) | 12 weeks
  The total distance walked in 6 minutes will be measured in meters
Physiological Outcome - handgrip | 12 weeks
  Handgrip will be measured in both the left and right hand. Two trials will be conducted on each side and the highest score will be used. Handgrip is measured in kg.
Physiological outcome - timed sit-to-stand | 12 weeks
  Time, is seconds, required to move from a seated to a standing position will be recorded.
Physiological Outcome - one legged stance/balance | 12 weeks
  Participants will be asked to stand on one leg with no support for as long as they can up to a maximum of 45 seconds. Trials will be conducted on the right and left side and time will be recorded in seconds.
Physiological Outcome - sit-and-reach | 12 weeks
  Hamstring flexibility will be measured in centimeters.
Physiological Outcome - shoulder flexibility | 12 weeks
  Shoulder flexibility will be measured in degrees
Daily steps | 12 weeks
  Total number of daily steps will be recorded using a pedometer.
Functional Assessment of Cancer therapy General (FACT-G) | 12 weeks
  The FACT-G is used to assess quality of life. It is a 27 item compilation of questions dived in four primary quality of life domains: 1) physical well-being; 2) social/family well-being; 3) emotional well-being; and 4) functional well-being.
Physical Activity Behaviour | 12 weeks
  The Godin Leisure Time Exercise Questionnaire will be used to assess physical activity and sedentary behaviour.
Sleep Quality | 12 weeks
  Sleep quality will be assessed using the Pittsburgh sleep quality index.
Depression Anxiety Stress Scales (DASS) | 12 weeks
  The depression anxiety stress scales consists of a list of 42 symptoms associated with depression, anxiety or stress. The participant is asked score the severity of the symptom over the past week on a 4 point scale.
Fatigue | 12-weeks
  The functional assessment of chronic illness therapy-fatigue (FACIT-F), which is a 13-item scale, will be used to assess participant levels of fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- QEII Health Sciences Centre (Dickson Bldg), Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No